CLINICAL TRIAL: NCT03230682
Title: Eealy Improvement Predicts Antidepressants Response in Adults With Major Depression Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jianhui Fu, Department of Neurology, Huashan Hospital, Huashan Hospital
Other Study IDs: KY2017-01
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Major Depressive Disorder
Keywords: early improvement; antidepressants; major depression diorder; resting-state fMRI
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Antidepressive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- major depressive disorder
  Interventions: Drug: antidepressant

INTERVENTIONS:
Drug: antidepressant — regular one-drups treatment of selective serotonin reuptake inhibitor(SSRIs)

SUMMARY:
Early improvemrnt, decreased 20% in the 17 items of Hamilton Depression Rating Scale (HAMD-17) at the second week of the treatment of major depression disorder (MDD), can arguably predict the remission at the 12th week. Our observation study including 80 MDD patients will access resting-state function MRI to finding factors which infuencing early improvemrnt, respone and remission of antidepressants.

ELIGIBILITY:
Inclusion Criteria:

* right-handed; HAMD-17 more than 17; diagnosed with MDD by the Structured Clinical Interview for DSM-IV

Exclusion Criteria:

* patients diagnosed with other condition in DSM-IV Axis I; pregnency; Thyroid disease; Heart Disease

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The han nationality who living in Shanghai, Zhejiang Province and Jiangsu Province
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2017-07-25 (Estimated); Primary Completion 2018-06-11 (Estimated); Study Completion 2018-07-11 (Estimated)

PRIMARY OUTCOMES:
Early improvement | the second week of treatment
  obtain 20% decrease of HAMD-17

SECONDARY OUTCOMES:
Response | the 12th week of treatment
  obtain 50% decrease of HAMD-17

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Neurology, Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wagner S, Engel A, Engelmann J, Herzog D, Dreimuller N, Muller MB, Tadic A, Lieb K. Early improvement as a resilience signal predicting later remission to antidepressant treatment in patients with Major Depressive Disorder: Systematic review and meta-analysis. J Psychiatr Res. 2017 Nov;94:96-106. doi: 10.1016/j.jpsychires.2017.07.003. Epub 2017 Jul 4. PMID 28697423
- [Result] Szegedi A, Jansen WT, van Willigenburg AP, van der Meulen E, Stassen HH, Thase ME. Early improvement in the first 2 weeks as a predictor of treatment outcome in patients with major depressive disorder: a meta-analysis including 6562 patients. J Clin Psychiatry. 2009 Mar;70(3):344-53. doi: 10.4088/jcp.07m03780. Epub 2009 Feb 24. PMID 19254516